CLINICAL TRIAL: NCT01094015
Title: Lidocaine-Prilocaine (EMLA) Cream as Analgesia in Hysteroscopy Practice: a Prospective Randomized Clinical Trial
Brief Title: Lidocaine-Prilocaine (EMLA) Cream as Analgesia in Hysteroscopy Practice
Acronym: HISTEROS-07
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Baldomero Arnau Rivera, Department of Gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HISTEROS-07
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2006-03

CONDITIONS: Pain
Keywords: hysteroscopy; local anaesthetic; pain relief; gynecological pathology
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine-Prilocaine cream (Active Comparator)
  Interventions: Drug: lidocaine-prilocaine cream
- placebo (Placebo Comparator)
  Interventions: Other: gel application for the transmission of ultrasound

INTERVENTIONS:
Drug: lidocaine-prilocaine cream — Implementation of 3 cm of lidocaine-prilocaine in the endocervical canal, 10 minutes before the intervention with a syringe without needle 5ml. Application, with a swab of the anesthetic cream ectocervix level.
  Other Names: EMLA
  Arms: Lidocaine-Prilocaine cream
Other: gel application for the transmission of ultrasound — 3 cm of gel application for the transmission of ultrasound into the endocervical canal 10 minutes before surgery, with a 5ml syringe without needle. Application, with a swab in gel ectocervix
  Other Names: Transonic-Gel
  Arms: placebo

SUMMARY:
The purpose of this study is to demonstrate that Lidocaine-Prilocaine cream decrease pain during hysteroscopy diagnostic practice.

ELIGIBILITY:
Inclusion Criteria:

* patients that he must perform a diagnostic hysteroscopy
* acceptance to participate in the study signed informed consent

Exclusion Criteria prerandomization:

* hypersensitivity or allergy to anesthetics
* refusal of the patient
* patients under age 18 and pregnant

Exclusion Criteria postrandomization:

* dropout
* unbearable pain that involves other analgesic measures
* allergic reactions to topical anesthetics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
pain reduction in the performance of hysteroscopy | after hysteroscopy and a month later
  decrease in pain immediately after the completion of hysteroscopy and one month after completion of the diagnostic test by an analogue pain scale

SECONDARY OUTCOMES:
sense of discomfort experience during the procedure | a month after hysteroscopy
  willingness to repeat the diagnostic technique

CONTACTS AND LOCATIONS:
Overall Officials: Baldomero Arnau, MD, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain